CLINICAL TRIAL: NCT02089971
Title: Muscle Mass and Function in Chinese Adults
Status: Completed | Type: Observational
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Other Study IDs: BL23
Record Dates: First submitted 2014-03-14; First posted 2014-03-18 (Estimated); Last update posted 2015-01-19 (Estimated); Status verified 2015-01

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Young Chinese adults: cross-sectional, observational study of community dwelling young Chinese adults

SUMMARY:
To describe the normal range of muscle mass and function in Chinese adults.

DETAILED DESCRIPTION:
The study objective is to setup a normal range of muscle mass and function in Chinese adults.

ELIGIBILITY:
Inclusion Criteria:

1. Young adult ages between 25 and 34 years, inclusively.
2. Adult is judged to be in good health as determined from his/her medical history as his/her self-report to the enrolling center personnel and as confirmed through a clinical examination by a physician.
3. Adult with BMI between 18.5 to 26.9.
4. Male or non-pregnant non-lactating female. Non-pregnant should be confirmed by urine pregnant test. And non-lactating is defined as postpartum more than 18 months.
5. Subject has voluntarily signed and dated an informed consent form, approved by an Independent Ethics Committee/Institutional Review Board (IEC/IRB) prior to any participation in the study.

Exclusion Criteria:

1. Subject who is heavy manual labor.
2. Subject who is professional or semi-professional athlete or game player.
3. Subject who is physical disabilities, such as loss of hand or foot or limbs or any physical disability which may affect the physical activities and affect the distribution of muscle mass by the opinion of the study physician.
4. Subject has known chronic diseases such as endocrine system diseases (including type 1 or type 2 diabetes mellitus, or hyperthyroidism or hypothyroidism), cardiovascular diseases, liver diseases, and renal diseases as self-report.
5. Subject who has active infection of TB, HIV and hepatitis as self-report.
6. Subject who currently experiencing diarrhea or anorexia within 7days prior to the enrollment.
7. Subject who has or plans for intensive physical activities 3 days prior to the scheduled BIA measurement.
8. Subject who is thyroid malfunction (as serum fT4 level and/or serum TSH level out of the reference range of the lab)
9. Subject has implanted electronic device, orthopedic metal implantations, such as pacemaker, cardiac defibrillator, or metal hip, metal knee joint, metal fracture internal fixation, etc.
10. Subject is drug addiction or alcohol addiction.
11. Subject is anemia (as blood hemoglobin level less than 120 g/L in males and 110 g/L in females).
12. Subject is malnourished by study physician's opinion
13. Subject has active cancers as self-report
14. Subject has lost or gained more than 5% of body weight in the past 3 months
15. Subject attends other clinical trials and is not approved by AN

Ages: 25 Years to 34 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Cross-sectional, observational study of young Chinese adults
Sampling Method: Non-Probability Sample
Enrollment: 412 (Actual)
Dates: Start 2014-03; Primary Completion 2014-10 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Total skeletal muscle mass | Test Visit 1 (~ Day 13)
  Dual X-ray Absorptiometry (DXA)

SECONDARY OUTCOMES:
Total body fat | Test Visit 1 (~ Day 13)
Total body fat free mass | Test Visit 1 (~ Day 13)
Total skeletal muscle mass | Test Visit 1 (~ Day 13)
  Bioelectrical Impedance Absorptiometry (BIA)

CONTACTS AND LOCATIONS:
Overall Officials: Xianfeng Zhao, MD, PhD, Study Chair — Abbott Nutrition China
Locations (2):
- China (2):
  - Peking Union Medical College Hospital, Beijing
  - Shanghai 6th People's Hospital, Shanghai